CLINICAL TRIAL: NCT07290504
Title: The Effect of Gradual Versus Intermittent Release of Tourniquet on Mean Arterial Blood Pressure in Hypertensive Patients Undergoing Upper Limb Orthopedic Surgeries: A Blinded Randomized Controlled Study
Brief Title: Gradual Versus Intermittent Release of Tourniquet Effect on MAP in Hypertensive Patients Undergoing Upper Limb Orthopedic Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Associate professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-77-2024/MSc
Record Dates: First submitted 2025-12-12; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hemodynamics
Keywords: Mean arterial pressure; Acid base; Tourniquet; Orthopedics; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: After completion of surgical procedure,tourniquet deflation will be performed by anesthesia technician into two ways according to the randomization number received in closed envelop with the patient file and blinded from the research anesthiologist: in gradual group (Ggroup) deflation by rate 50mmHg/ 30s untill complete release within 3 minutes .In intermittent group (Igroup) complete deflation will occur for 10 seconds, then reinflated for 50 seconds, repeating this cycle three times until complete release.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: After completion of surgical procedure, tourniquet deflation will be performed by anesthesia technician into two ways according to the randomization number received in closed envelop with the patient file and blinded from the research anesthiologist: in gradual group (Ggroup) deflation by rate 50mmHg/ 30s untill complete release within 3 minutes .In intermittent group (Igroup) complete deflation will occur for 10 seconds, then reinflated for 50 seconds, repeating this cycle three times until complete release.The researcher anesthesiologist who collects data, including hemodynamics and labs will be separated from the upper limb, tourniquet device, and the technician by surgical curtain to ensure full blinding of the deflation technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G group (Experimental): Gradual group (G group) deflation by rate 50mmHg/ 30s until complete release within 3 minutes
  Interventions: Device: Tourniquet deflation
- I group (Active Comparator): Intermittent group (I group) complete deflation will occur for 10 seconds, then reinflated for 50 seconds, repeating this cycle three times until complete release.
  Interventions: Device: Tourniquet deflation

INTERVENTIONS:
Device: Tourniquet deflation — Tourniquet deflation technique

SUMMARY:
In this clinical trial, the authors will compare two tourniquet deflation techniques and their clinical implications on hemodynamics and acid base parameters in hypertensive orthopedic patients undergoing upper limb surgeries under general anesthesia.

DETAILED DESCRIPTION:
General anesthesia will be induced using an injection of 1-1.5 mg/kg of propofol, 1-2 mic/kg of fentanyl, and 0.5 mg/kg of atracurium,with all doses to be titrated. An endotracheal tube will be inserted after 3 minutes of mask ventilation.

Anesthesia will be maintained using isoflurane (1%) and atracurium at a dosage of 0.1mg\kg every 20 minutes.

After endotracheal intubation, the patients will be mechanically ventilated with a 50% oxygen-air mixture, utilizing a tidal volume of 8 mL/kg based on ideal body weight at an inspiratory rate of 10-14 breaths per minute. Adjustments will be made to ensure that the end-tidal CO2 partial pressure (ETCO2) between 35 and 40 mmHg, with peak airway pressure kept below 30 mmHg.

The surgeon will start limb elevation, exsanguinating of blood and applying a double- cuffed tourniquet(zimmer A.T.S.3000) at the middle of the arm over cotton padding,with pressure ranging 200 mmHg according to the patient's blood pressure (50mmHg above systolic blood pressure).

After completion of surgical procedure,tourniquet deflation will be performed by anesthesia technician blinded to the study groups into two ways according to the randomization number received in closed envelop with the patient file and blinded from the research anesthiologist: in gradual group (G group) deflation by rate 50mmHg/ 30s untill complete release within 3 minutes .In intermittent group (I group) complete deflation will occur for 10 seconds, then reinflated for 50 seconds, repeating this cycle three times until complete release. If the surgery exceeded 2 hr, the intermittent technique for deflation will be used The researcher anesthesiologist who collects data, including hemodynamics and labs will be separated from the upper limb, tourniquet device, and the technician by surgical curtain to ensure full blinding of the deflation technique.

A bolus of lidocaine 1.5 mg\kg will be administered 10 minutes before tourniquet inflation will be used to attenuate the increase of blood pressure after tourniquet inflation.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients (controlled on medical treatment more than three months)
* Patients scheduled for upper limb orthopedic surgeries using a tourniquet for at least 30 min.
* BMI from 18.5 to 29.9

Exclusion Criteria:

* Patient refusal
* ASA physical status > II
* Multiple orthopedic surgeries
* Emergency surgeries
* Patient with relative contraindications for tourniquet use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean Arterial Pressure | 5 minutes
  The decrease in MAP (more than 25% compared to baseline) 5 minues after deflation.

SECONDARY OUTCOMES:
Acid base status | 5 minutes
  Acid base status
Lactate | 30 minutes
  Lactate level
Potassium level | 30 minutes
  Potassium level

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No